CLINICAL TRIAL: NCT06778798
Title: Pain Reduction of an Oral Gabapentin and Median Nerve Neural Mobilization Combined Treatment Compared to Only Oral Gabapentin in Subjects Who Suffer Carpal Tunnel Syndrome
Brief Title: Gabapentin and Neural Mobilization Pain Reduction Effect Compared to Only Gabapentine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Francisco Unda Solano, Biomedicine Doctorate Program Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CE0072015-02-06
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Gabapentin; Median nerve neural mobilization; Pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Median nerve neural mobilization and oral gabapentin (Experimental): Median nerve neural mobilization, non pharmaceutical, non invasive, physiotherapy technique; which consists of a passive and repetitive upper limb movement that seeks to induce median nerve gliding and incursions against surrounding connective tissue. Subjects will be treated 5 days per week during a total time lapse of 2 weeks. This arm will also receive a Gabapentin Oral capsule pharmaceutical treatment. Participants will be treated with a maximum of 600 mg per day, subdivided in 2 intakes of 300 mg each 12 hours during a time lapse of 2 weeks.
  Interventions: Combination Product: Median nerve neural mobilization and oral gabapentin
- Gabapentin (Active Comparator): Gabapentin Oral capsule pharmaceutical treatment. Participants will be treated with a maximum of 600 mg per day, subdivided in 2 intakes of 300 mg each 12 hours during a time lapse of 2 weeks.
  Interventions: Drug: Gabapentin 300mg

INTERVENTIONS:
Combination Product: Median nerve neural mobilization and oral gabapentin — Manual therapy maneuver performed in the upper limb combined with gabapentin oral capsules.
  Arms: Median nerve neural mobilization and oral gabapentin
Drug: Gabapentin 300mg — Gabapentin oral capsules
  Other Names: Neurontin
  Arms: Gabapentin

SUMMARY:
In the present investigation the pain reduction effects of a physiotherapy technique combined with pharmaceutical gabapentin treatment will be compared to those produced by gabapentin (only) treatment, in subjects who suffer the signs and symptoms of carpal tunnel syndrome.

DETAILED DESCRIPTION:
The present randomized clinical trial will perform a comparison of the pain reduction effects produced by the application of a non invasive and non pharmacological median nerve neural mobilization (physiotherapy treatment) combined with a pharmaceutical oral gabapentin treatment, to those effects produced by a gabapentin (only) treatment. Additionally, effects over the functionality of the affected upper limb will be evaluated and compared. Subjects will be invited to participate and randomly allocated to 2 different groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be medically diagnosed with unilateral carpal tunnel syndrome (with confirmative electrodiagnostic findings).
* Full understanding of written and spoken Spanish (language).
* Participants must freely consent to participate.
* The presence of positive Phalen and Tinel signs.
* The presence of carpal tunnel syndrome signs and symptoms

Exclusion Criteria:

* The lack to meet inclusion criterions, the presence of cognitive impairment, tumors, cancer, recent (affected) upper limb surgery or trauma, pregnancy, metabolic neuropathy, obesity (body mass index over 30), participants who are not employed, deformities of the (affected) upper limb, recent skin injuries or infections (in the affected upper limb), autoimmune inflammatory conditions or flu type symptoms, allergy to gabapentin, allergy to ibuprofen arginine, and also: participants must not be (during the present investigation) under any type of pain reducing treatment (conservative, homeopathic, invasive or not invasive)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Distal upper limb pain | Through study completion, an average of 2 weeks. Changes from baseline (measured immediately before the application of the first treatment) and 40 minutes after the application of the last treatment.
  Assessed through the visual analog scale (VAS). The VAS is a psychometric response scale. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. The VAS is the most frequently used method to assess pain intensity. The scale will be displayed as a horizontal 10-cm line labelled at each end by descriptors such as 'no pain' (the minimum and best outcome possible) and 'worse pain ever' (maximum and worst outcome possible). The participant will mark the line to indicate pain severity and it is simply quantified by measuring the distance in centimeters from 0 (no pain) to the patient's marked rating.

SECONDARY OUTCOMES:
Upper limb function | Through study completion, an average of 2 weeks.Changes from baseline (measured immediately before the application of the first treatment) at 40 minutes after the application of the last treatment.]
  Assessed through the QuickDASH questionary, which is a shortened version of the 30-item DASH (Disabilities of the Arm, Shoulder and Hand) instrument.The instrument administered to the participants will be a self-report questionnaire, that will rate the difficulty and interference of daily life on a 5 point Likert scale. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability).
Work Status at baseline | Measured immediately before the application of the first treatment
  This measure is performed through the employed participant (full-time or part-time) answering in a dichotomous manner (yes or no) the question: "Do you currently work?"
Work Status post treatment | Measured immediatly after the application of the last treatment.
  This measure is performed through the employed participant (full-time or part-time) answering in a dichotomous manner (yes or no) the question: "Do you currently work?"
Change in Work Task (Job Type) | Measured immediatly after the application of the last treatment.
  This measure is performed through the employed participant (full-time or part-time) answering in a dichotomous manner (yes or no) the question: "Did you change your job type or task?"
Tampa Scale for Kinesiophobia-17 (TSK-17) | Changes from baseline (measured immediately before the application of the first treatment), and at 60 minutes after the application of the last treatment.
  The Tampa Scale for Kinesiophobia-17 (TSK-17) is a 17-item questionnaire designed to assess the fear of movement and re-injury (kinesiophobia). Items are rated on a 4-point Likert scale (ranging from "strongly disagree" to "strongly agree"), yielding a total score that reflects the severity of pain-related fear avoidance beliefs. It's a widely used and vailidaded clinical and research instrument. The standard total score range for the Tampa Scale for Kinesiophobia (TSK-17) is 17 to 68. It is calculated by summing 17 items, each scored 1-4, with four items reverse-scored. Higher scores indicate greater fear of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Unda, PhD, Principal Investigator
Locations (1):
- Ciudad Hospitalaria Enrique Tejera, Valencia, Carabobo, Venezuela

IPD SHARING:
Plan to Share IPD: No